CLINICAL TRIAL: NCT02247310
Title: BETAEVAL_Global- The New BETACONNECT® Auto-injector: Adherence and EVALuation of MS Patients Treated With Betaferon®
Brief Title: BETAEVAL Global - The New BETACONNECT Auto-injector : Adherence and EVALuation of Multiple Sclerosis Patients Treated With Betaferon
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17591; BF1401 (Other: Company Internal)
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with the diagnosis of relapsing remitting multiple sclerosis or a clinically isolated syndrome and be on treatment with Betaferon using the BETACONNECT auto-injector device.
  Interventions: Drug: Interferon beta-1b (Betaferon®, BAY 86-5046); Device: BETACONNECT

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon®, BAY 86-5046) — Patients will be treated with Betaferon
Device: BETACONNECT — Auto-injector device to support the injection of Betaferon

SUMMARY:
Considering the significance of an early and consequent Multiple Sclerosis (MS) treatment as well as the challenge to achieve high adherence to treatment, evaluating the benefits of any new measure to improve adherence is important. The data storage capabilities of the BETACONNECT device, including the automated recording of injections, will facilitate the collection of reliable data on patient's injection behavior and adherence, which should be unaffected by recall bias or reporting bias.

To better understand the utilities of the new BETACONNECT device and characterize its contribution to adherence, we plan to prospectively follow-up MS patients using this device for 24 weeks. The study will take place in a real-life setting in Neurology centers across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of relapsing remitting multiple sclerosis or a clinically isolated syndrome.
* Patients must be on treatment with Betaferon or the decision to treat a patient with Betaferon has been made by the attending physician.
* Patient and attending physicians must have agreed on the usage of the BETACONNECT auto-injector device.
* Written informed consent must be obtained.

Exclusion Criteria:

* Patients receiving any other disease modifying drug.
* Contraindications of Betaferon described in the Summary of Product Characteristics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with relapsing remitting multiple sclerosis (RRMS) or patients with a clinically isolated syndrome (CIS) who are treated with Betaferon or will be treated with Betaferon® according to the attending physician's decision and for whom the patient and the physician have agreed to use the BETACONNECT device.
  The study will be conducted in neurological centers and neurology departments specialized in the treatment of Multiple Sclerosis patients.
Sampling Method: Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Adherence to therapy at the final visit. | Up to 24 weeks

SECONDARY OUTCOMES:
Satisfaction with and evaluation of the BETACONNECT auto-injector | At baseline,4 weeks,12 weeks and 24 weeks
  Satisfaction with and evaluation of the BETACONNECT auto-injector will be recorded with the patient questionnaire
Injection site pain and prophylactic analgesic use | At baseline,4 weeks,12 weeks and 24 weeks
  Injection site pain and prophylactic analgesic use will be recorded with the patient questionnaire
Health related quality of life | At baseline,12 weeks and 24 weeks
  Health related quality of life will be measured with the self-administered Functional Assessment of Multiple Sclerosis (FAMS) questionnaire.
Anxiety | At baseline,12 weeks and 24 weeks
  Anxiety will be measured with the self-administered Hospital anxiety and depression scale (HADS).
Depression | At baseline,12 weeks and 24 weeks
  Depression will be measured with the self-administered Center for Epidemiologic Studies Depression Scale (CES-D).
Fatigue | At baseline,12 weeks and 24 weeks
  Fatigue will be measured with the self-administered Fatigue Scale for Motor and Cognitive functions (FSMC).
Cognition | At baseline,12 weeks and 24 weeks
  Cognition will be measured by the HCP with the Symbol Digit Modalities Test (SDMT).
Local skin reactions | At baseline,4 weeks,12 weeks and 24 weeks
  Local skin reactions will be recorded by HCP evaluation (local inspection).
Injection-related specifics | At 4 weeks,12 weeks and 24 weeks
  Injection-related specifics such as injection date, time, and speed will be recorded by the BETACONNECT device

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Bosnia and Herzegovina
- Many Locations, Croatia
- Many Locations, Czechia
- Many Locations, France
- Many Locations, Greece
- Many Locations, Hungary
- Many Locations, Italy
- Many Locations, Spain
- Many Locations, Switzerland